CLINICAL TRIAL: NCT01796210
Title: Prediction of Hemodynamic Reactivity During Suspension Laryngoscopy Using Analgesia/Nociception Index (ANI): an Observational Study
Brief Title: Prediction of Hemodynamic Reactivity During Suspension Laryngoscopy Using Analgesia/Nociception Index (ANI)
Status: Completed | Type: Observational
Sponsor: Emmanuel Boselli (Other)
Responsible Party: Sponsor-Investigator, Emmanuel Boselli, MD, PhD, Hôpital Edouard Herriot
Organization: Hôpital Edouard Herriot (Other)
Other Study IDs: CPP 2012-046B
Record Dates: First submitted 2013-02-18; First posted 2013-02-21 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Anesthesia
Keywords: Analgesia/nociception index; Bispectral index; Propofol; Remifentanil; Suspension laryngoscopy; Endoscopy; Ear-nose-throat
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to evaluate the performance of Analgesia/Nociception Index for the prediction of hemodynamic reactivity in adult patients undergoing suspension laryngoscopy on general anesthesia.

DETAILED DESCRIPTION:
Measurement of analgesia/nociception index at different time points during procedure and assessment of analgesia/nociception index to predict hemodynamic reactivity by building receiver observer's characteristic curve.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Suspension laryngoscopy for diagnostic or therapeutic purposes
* Total intravenous anesthesia using propofol and remifentanil

Exclusion Criteria:

* age <18 yrs or >75 yrs
* arrythmia
* administration of anticholinergic drugs or neuromuscular blockade reversal in the 20 previous minutes
* psychiatric diseases
* autonomic nervous system disorders (epilepsy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients underoing suspension laryngoscopy performed on general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in heart rate and/or systolic blood pressure by more than 20% within 5 minutes | Before induction of anesthesia, 1 min after beginning of procedure, at steady-state anesthesia during procedure (an expected average of 10 min) and at arousal from general anesthesia in the end of procedure (an expected average of 20 min)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Boselli, MD, PhD, Study Director — Hôpital Édouard Herriot, HCL
Locations (1):
- Hôpital Édouard Herriot, HCL, Lyon, Rhône, France